CLINICAL TRIAL: NCT05718765
Title: The Effect of Physical ACtivity Enhancement Scheme (PACES) on Physical Outcomes in Hemodialysis Patients
Brief Title: The Effect of Physical ACtivity Enhancement Scheme (PACES) in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Mei Huang, Principal Investigator, Xi'an Jiaotong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022SF-077
Record Dates: First submitted 2022-12-24; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Kidney Failure, Chronic; Exercise; Physical Activity; Renal Dialysis
Keywords: End-Stage Renal Disease; Exercise; Physical Activity; Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care with sham intervention (Sham Comparator): Patients in the control group received usual care with sham exercise.
  Interventions: Other: Usual care with sham intervention
- PACES intervention (Experimental): PACES includes an exercise perception intervention and an exercise intervention, which lasts for 12 weeks and is carried out simultaneously.
  Interventions: Behavioral: PACES intervention

INTERVENTIONS:
Behavioral: PACES intervention — The exercise perception intervention program is divided into three stage, and every four weeks is a stage. The theme of the first stage is to make the patient have the intention to exercise. The theme of the second stage is to provide effective support for the patient, so that the patient can take the initiative to start exercise. The theme of the third stage is to enable patients to keep exercising.
  The exercise intervention is a 12-week progressive intradialytic combined cycling exercise which proceed in the first HD 2 hours for safety. Each session consisted of a 5-minute warm-up, cool-down and 30-minute cycling at a Rating of Perceived Exertion (RPE) of 12-14. The machine has two exercise types including aerobic exercise and resistance exercise. Every four weeks is divided into a stage. And the time of aerobic exercise and resistance exercise were personally adjusted per stage to maintain the personalized target RPE.
  Arms: PACES intervention
Other: Usual care with sham intervention — Patients in the control group received usual care and were advised to do sham exercise such as stretch legs and arms about 15 minutes during the first 2 hemodialysis hours.
  Arms: Usual care with sham intervention

SUMMARY:
Hemodialysis is the most commonly used renal replacement therapy for end-stage renal disease (ESRD) patients. At present, more than 553,000 ESRD patients in China are receiving hemodialysis treatment, but the long-term survival rate is low, and the annual mortality rate is as high as 18%. This is significantly related to lower physical activity in hemodialysis patients. Physical inactivity can lead to the decline of cardiopulmonary function and muscle function, the aggravation of daily life restriction and the increased risk of death. The National Kidney Foundation Disease Outcomes Quality Initiative (K/DOQI) recommends physical activity as cornerstone of ESRD rehabilitation. But hemodialysis patients are still living in a physical inactivity state. In the early stage of this study, the Physical Activity Enhancement Scheme (PACES) was developed for hemodialysis patients, that is, taking spaces as the core of physical activity investigation, and encouraging patients to start to improve physical activity. The PACES has been registered on the ClinicalTrials.gov before (number: NCT05189795).

The investigators now plan to evaluate the impact of PACES on physical activity of hemodialysis patients through clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* adult (age≥18) with stable ESRD;
* receiving≥3 months HD;
* receiving HD more than 5 times every two weeks;
* volunteer for participating in this investigation.

Exclusion Criteria:

* are unable to do walk on one's own (severe musculoskeletal pain at rest or with minimal activity precluding walking or stationary cycling; unable to sit, stand or walk unassisted, walking devices such as cane or walker allowed);
* have shortness of breath at rest or with activities of daily living (NYHA Class IV);
* have mental disease, disturbance of consciousness and couldn't cooperate with this investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
daily steps (paces) | Change from daily steps at 12 weeks.
  OMRON electronic pedometer (HJ-321) records the participants' daily steps. Participants are instructed to wear the pedometer on their waist for 7 days, and the pedometer is removed only during rest, bathing and swimming.
The Human Activity Profile (HAP) | Change from HAP 12 weeks.
  HAP is a questionnaire designed to assess general physical activity. It consists of a list of 94 activities ranked in ascending order of level of energy required to perform each activity. Two scores are available from the HAP: a maximum activity score (MAS), reflective of the most taxing activity a respondent is still performing and an adjusted activity score (AAS), reflective of the respondent's daily activity level. The MAS is the number of the highest ranked activity the respondent is still performing. The AAS is calculated by subtracting from the MAS the number of activities that the respondent has stopped performing that rank below the participants' most metabolically intense activity. The minimum and maximum values of MAS and AAS are 0 and 94 respectively. The higher the score, the stronger the physical activity of the patient.

SECONDARY OUTCOMES:
Dialysis Patient-perceived Exercise Benefits and Barriers Scale (DPEBBS) | DPEBBS is measured at baseline (before intervention) and after 12 weeks of intervention.
  The 24-item DPEBBS is used to evaluate participants' perceived benefits and barriers to exercise. The scale consisted of 24 items and 2 open questions, including 12 items of exercise benefits and 12 items of exercise barriers. Total scores ranged from 24 to 96. The higher the score, the more exercise benefits the patients experienced and the fewer factors that prevented them from exercise.
Self-efficacy for exercise scale (SEE) | SEE is measured at baseline (before intervention) and after 12 weeks of intervention.
  SEE is used to identify the participants' confidence in their ability to exercise, which is a major determinant in the success of changing behavior. The score ranges from 0 to 100, and the higher the score, the higher the level of self-efficacy.
Social support Rating Scale (SSRS) | SSRS is measured at baseline (before intervention) and after 12 weeks of intervention.
  Participants' social support status is measured by the SSRS. The scale has 10 items, including 3 aspects, objective support, subjective support and utilization of social support. The total score is the sum of points for each item. The higher the score is, the higher the degree of social support is. The scale scores range from 12 to 66, with ≤22 being low, 23 to 44 medium, and 45 to 66 high.
Stage of Change Questionnaire | The questionnaire is measured at baseline (before intervention) and after 12 weeks of intervention.
  The questionnaire identifies the participants' state of readiness to adopt a more active lifestyle according to the Health Action Process Approach. The higher the stage, the better the readiness of the participants.
Kidney Disease Quality of Life (KDQOL-36) | KDQOL-36 is measured at baseline (before intervention) and after 12 weeks of intervention.
  KDQOL-36, consisted of the 12-item Short Form Health Survey (SF-12) including the physical component summary (PCS) and the mental component summary (MCS) and 24 disease-specific items which entail 3 subscales: the symptom and problems list, the burden of kidney disease, and the effects of kidney disease, is to evaluate patients' QoL. Scores of each dimension range from 0 to 100 and higher scores represent better QoL.
Glomerular filtration rate (GFR) | GFR is measured at baseline (before intervention) and after 12 weeks of intervention.
  GFR is estimated by the using the CKD-EPI creatinine equation.
Serum levels of IL-6 | Serum levels of IL-6 is measured at baseline (before intervention) and after 12 weeks of intervention.
  Serum levels of IL-6 is measured using immunoassay kit (DuoSet ELISA Development, R&D Systems, Inc., USA). Blood samples are drawn after an overnight fast of at least 12 hour. The last blood collection will be performed 48 h after the last exercise session, to avoid acute effects of the exercise influencing inflammatory and oxidative stress markers. These methods will follow the manufacturer's recommendations.
C-reactive protein (CRP) | CRP is measured at baseline (before intervention) and after 12 weeks of intervention.
  CRP is evaluated as an index of catabolism and systemic inflammation using a high-sensitivity assay.
Serum creatinine | Serum creatinine is measured at baseline (before intervention) and after 12 weeks of intervention.
  Serum creatinine is evaluated as an index of catabolism and systemic inflammation.
sit-to-stand tests 10 (STS-10) | STS-10 is measured at baseline (before intervention) and after 12 weeks of intervention.
  The sit-to-stand tests 10(STS-10) is a test that assesses the capacity to stand up from a chair. The STS-10 is calculated as the total time needed to complete 10 repetitions of standing up and sitting down again.
sit-to-stand tests 60 (STS-60) | STS-60 is measured at baseline (before intervention) and after 12 weeks of intervention.
  The sit-to-stand tests 60 (STS-60) is a test that assesses the capacity to stand up from a chair. The STS-60 registers the repetitions performed in 60 seconds.
Six-minute walk test (6MWT) | 6MWT is measured at baseline (before intervention) and after 12 weeks of intervention.
  6MWT is commonly used to assess walking capacity in patients with chronic diseases, including Chronic Kidney Disease (CKD) patients.
Ejection fraction | Ejection fraction is measured at baseline (before intervention) and after 12 weeks of intervention.
  Transthoracic echocardiography is performed using a Vivid E95 ultrasound system (General Electric, Frankfurt, Germany) equipped with a multifrequency transducer and 4D imaging analysis software. Normative ultrasound images were obtained by use of a 3.5-MHz phased array probe, placed on the third or fourth left intercostal space and Apical region. Connect electrocardiogram (ECG) for each subject to ensure standardization of image acquisition and data calculation to obtain ejection fraction. Data were analyzed and interpreted by one experienced echocardiographer who was blinded to treatment status and imaging sequence. To minimize the effect of variations in fluid volume in hemodialysis patients, studies were performed 18-24 h after a hemodialysis session.
Left ventricular mass index | Left ventricular mass index is measured at baseline (before intervention) and after 12 weeks of intervention.
  Left ventricular mass is calculated from M-mode images, according to the guidelines of the American Society of Echocardiography. The left ventricular mass index is obtained by dividing by the formula of body surface area.
Left ventricular volume index | Left ventricular volume index is measured at baseline (before intervention) and after 12 weeks of intervention.
  Left ventricular volume is calculated from M-mode images, according to the guidelines of the American Society of Echocardiography. The left ventricular volume index is obtained by dividing by the formula of body surface area. index is obtained by dividing by the formula of body surface area.

CONTACTS AND LOCATIONS:
Locations (1):
- Nursing School of the Air Force Medical University, Xi'an, Shaan XI, China